CLINICAL TRIAL: NCT04980430
Title: Evaluating Community Interest in Virtual Reality Vision Screening Technology
Brief Title: Community Interest in Vision Screening Technology
Acronym: RTS2
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, James Chelnis, Assistant Clinical Professor, Icahn School of Medicine at Mount Sinai
Other Study IDs: Study-20-00358
Record Dates: First submitted 2021-07-18; First posted 2021-07-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Ophthalmology; Vision Screening
Keywords: Ophthalmology; Virtual Reality; Community; Vision

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Primary Care and Ophthalmology clinic patients: Participants will be recruited from primary care and ophthalmology clinics in New York City
  Interventions: Device: Virtual Reality

INTERVENTIONS:
Device: Virtual Reality — Virtual Reality Demonstration

SUMMARY:
Virtual reality (VR) is a relatively new, emerging field within healthcare. Studies have analyzed public perceptions of virtual reality in healthcare using social media, but few have actually demonstrated and educated these modalities to communities. Because vision care can be costly and inaccessible, especially in communities with few physicians, this study aims to evaluate whether communities would be open to new technology. For example, it has been determined that 80% of vision loss is preventable with adequate screening technology, a key factor in ameliorating the economic and emotional burden of eye disease. Therefore, through demonstrations and educational presentations by medical students, gaps in understanding perceptions, willingness to adopt, and general demographics of those seeking better eye care will be understood.

DETAILED DESCRIPTION:
This study is critical to show healthcare leaders that communities seek new, lower cost, and more accessible technologies for vision care. This study will also be used to expand use of the technology in other communities and prove a use case for it. Ultimately, this can help benefit communities to ensure that all are receiving proper vision care and to address common conditions in a timely manner.

If participants agree to participate, individuals will be educated about vision care and the use of virtual reality technology by a medical student or trained volunteer using a VR headset. This entire process will take about 5 minutes. Participants will be allowed to take breaks and medical students and/or volunteers will be nearby to answer any questions they may have throughout the study. There will be no results given to patients during the study nor will they be advised to use any information to inform future healthcare decisions. The purpose of the study is demonstrative.

After the demonstration, a survey will be given to each participant about their experience with the VR technology along with demographic information. This will be kept confidential and will only be accessed by those approved. The survey will take approximately 5 minutes. In addition, we will offer educational materials on the conditions that the vision tests are used to screen for.

ELIGIBILITY:
Inclusion Criteria:

* Males and females of any race
* At least 18 years of age
* Participants must be able to understand and provide verbal and written consent. Only participants who undergo the demonstration of the technology and consent to the study after full explanation will be included in research.

Exclusion Criteria:

- People who have undergone intraocular surgery less than six months ago, and potential contraindication for visual field test that include anxiety disorder, pregnancy, seizure disorder, cardiac pacemaker or another implantable device, severe vertigo or balance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from primary care and ophthalmology clinics in New York City. Participants can schedule a time to participate in the study on their own or may be recruited by a student at their appointment.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
Virtual Reality Assessment | Day 1
  Participant assessment of VR technology. Items scored on a likert-scale format from 1 (strongly disagree) to 5 (strongly agree). Full scale from 13 to 65, with higher score indicating more favorable responses.

SECONDARY OUTCOMES:
Demographics Assessment | Day 1
  Survey to evaluate participant demographics and vision care needs. This is not a scored or scaled survey.

CONTACTS AND LOCATIONS:
Overall Officials: James Chelnis, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Ophthalmology Faculty Practice Associates, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Immediately following publication. No end date.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ('learned intermediary') identified for this purpose. Any purpose. Data available on specific request and will be shared securely as CSV